CLINICAL TRIAL: NCT05165017
Title: Randomized Double Blind Placebo Controlled Study of the Safety & Efficacy of Therapeutic Treatment With AlloRx Stem Cells® in Patients With Pitt Hopkins Syndrome (Phase 1/2 Study)
Brief Title: Safety & Efficacy of AlloRx SC® in PTHS Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vitro Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALLORX-PTHS
Record Dates: First submitted 2021-10-29; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Pitt Hopkins Syndrome
MeSH Terms: conditions — Pitt-Hopkins syndrome

STUDY DESIGN:
Intervention Model Description: Randomized Placebo Controlled Double Blinded
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention Arm 1 (Active Comparator): AlloRx Stem Cells IV infusion treatment
  Interventions: Biological: AlloRx Stem Cells®
- Intervention Arm 2 (Placebo Comparator): IV infusion of normal saline
  Interventions: Other: Placebo control

INTERVENTIONS:
Biological: AlloRx Stem Cells® — Umbilical cord-derived allogeneic mesenchymal stem cells
  Arms: Intervention Arm 1
Other: Placebo control — Placebo infusion without mesenchymal stem cells
  Arms: Intervention Arm 2

SUMMARY:
This study will evaluate the safety of AlloRx Stem Cells® in subjects with Pitt Hopkins syndrome ages 2-45 with a molecularly confirmed pathogenic mutation in TCF4 or 18q deletion including TCF4. Participants will receive mesenchymal stem cells infusions every 3 months for a year with completion of outcome measures to assess the efficacy of the product.

DETAILED DESCRIPTION:
This is a phase 1/2, randomized placebo controlled double blinded standard dose study to evaluate the safety and tolerability of AlloRx® stem cells in pediatric patients with a confirmed diagnosis of a TCF4 mutation consistent with haploinsufficiency causing PTHS. Approximately 26 patients (male and female) ages ≥ 2 and≤ 45 years of age with a genetically confirmed diagnosis of Pitt-Hopkins syndrome caused by molecular findings consistent with a pathogenic mutation in the gene TCF4. Written informed consent will be obtained from the patient's parent or legal guardian/ authorized representative (LAR) prior to participation in the study. The study includes screening, baseline, treatment and safety follow up periods. The procedure for intravenous administration is performed under the supervision of clinician with experience caring for patients with PTHS.

Each patient will remain inpatient for at least 24 hours after the initial dose of AlloRx, for frequent vital sign monitoring, electrocardiogram (ECG), blood and urine safety tests, and neurologic assessments. Investigators will work closely with the parent/legal guardian to ensure that any signs of discomfort/distress are immediately communicated to study staff. For the administration of the initial dose of study drug in each study cohort, patients will be dosed in a sequential fashion with no more than one patient receiving their first dose of study drug on the same day.

An independent data DSMB will review all safety and laboratory data throughout the study on a periodic basis and ad hoc should an SAE occur. The DSMB will also review all available safety data when all patients have received 2 doses of AlloRx and have had at least two weeks of follow-up in order to determine if it is safe to dose the next patient.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from parent(s) or legal guardian(s)/authorized representative(s) (LAR)
* Documented genetic confirmation of mutation in TCF4, with clinical diagnosis of Pitt Hopkins Syndrome (PTHS)
* Stable seizure control (defined as clinically stable with no changes in antiepileptic medications or use of rescue medication over the prior 1 month before the screening visit, other than weight associated dose adjustments)
* Normal renal function with serum creatinine and spot urine protein within normal limits
* Willing and able to comply with scheduled visits, drug administration plan, laboratory tests, study restrictions, and all study procedures, including intravenous infusion

Exclusion Criteria:

* Any change in medications or diet/supplements intended to treat symptoms of PTHS (e.g., sleeping aids, supplements, cannabidiol products) over the prior 3 months before screening
* Inability to ambulate independently or with an assistive device or caregiver handhold
* Any bleeding or platelet disorder
* Any clinically significant (CS) cardiovascular, endocrine, hepatic, renal, pulmonary, gastrointestinal, neurologic, malignant, metabolic, psychiatric, or other condition that, in the judgment of the Investigator, will pose a safety risk, make the patient unsuitable for participation in, and/or unable to complete the study procedures
* Any laboratory abnormality, that, in the Investigator's opinion, could adversely affect the safety of the patient, make it unlikely that the course of treatment or follow up would be completed, or impair the assessment of study result
* Known positive for hepatitis B virus, hepatitis C virus, or human immunodeficiency virus (HIV). Patient is pregnant or lactating
* Usage of drugs that increase the risk of bleeding (e.g., heparin, low molecular weight heparin, platelet inhibitors).
* Use of any investigational oligonucleotide and any investigational drugs in the past 6 months
* Any prior use of gene therapy

Ages: 2 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events improvement) in one or more areas of ailments related to PTHS | Change from baseline to day 456 (end of study)
  Collection of all adverse events (AEs)
Safety: Incidence of serious adverse events | Change from baseline to day 456 (end of study)
  Collection of all serious adverse events

SECONDARY OUTCOMES:
Change in motor function in individuals with PTHS | Change from baseline to day 456 (end of study)
  Ambulation measures by video and wearable device
Change in communication abilities in individuals with PTHS. | Change from baseline to day 456 (end of study)
  Observer-Reported Communication Ability Measure (ORCA)
Change in sleep habits | Change from baseline to day 456 (end of study)
  Sleep diary
Change in gastrointestinal health | Change from baseline to day 456 (end of study)
  Gastrointestinal Health Questionnaire
Change in breath holding spells | Change from baseline to day 456 (end of study)
  Diary of breath holding spells
Change in cognition | Change from baseline to day 456 (end of study)
  Bayley Scales of Infant Development (BSID-4)
Change in adaptive function | Change from baseline to day 456 (end of study)
  Vineland Adaptive Behavioral Scale-3
Change in autistic features | Change from baseline to day 456 (end of study)
  Childhood Autism Rating Scale (CARS)
Change in parent assessment of quality of life | Change from baseline to day 456 (end of study)
  Pediatric Quality of Life Questionnaire
Change in global clinical status | Change from baseline to day 456 (end of study)
  PTHS-specific Clinical Global Impression Scale

IPD SHARING:
Plan to Share IPD: No